CLINICAL TRIAL: NCT04360538
Title: Long Term Outcomes of Patients With COVID-19
Acronym: COVID19 LTFU
Status: Active, not recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0538
Record Dates: First submitted 2020-04-16; First posted 2020-04-24 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Critical Illness; Corona Virus Infection; Respiratory Failure; Covid-19
Keywords: long term outcomes; mechanical ventilation; noninvasive ventilation
MeSH Terms: conditions — Critical Illness; Coronavirus Infections; Respiratory Insufficiency; COVID-19 | interventions — Quality of Life; 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID19 positive: ICU patients coronavirus positive
  Interventions: Other: Quality of Life; Other: Impact Event Score; Other: Hospital anxiety and depression scale
- non-COVID19: ICU patients without coronavirus
  Interventions: Other: Quality of Life

INTERVENTIONS:
Other: Quality of Life — Physical disability assessment tool
  Other Names: SF-36
Other: Impact Event Score — Psychological Sequelae assessment tool
  Other Names: IES-R
  Groups: COVID19 positive
Other: Hospital anxiety and depression scale — Psychological Sequelae assessment tool
  Groups: COVID19 positive

SUMMARY:
The investigators hypothesize that those with respiratory failure due to COVID-19 will have different burdens of mental and physical disability than those with respiratory failure who do not have COVID-19. Detecting these potential differences will lay an important foundation for treating long term sequelae of respiratory failure in these two cohorts.

DETAILED DESCRIPTION:
The aim of this proposal to is to understand the extent and degree of physical disability, psychological sequelae, and cognitive dysfunction survivors of COVID-19 related critical illness will have upon hospital discharge, 6 months, and up to one year post discharge. These outcomes of interest will be evaluated prospectively. The investigators will perform these measures in Covid-19 patients with respiratory failure and compare them to non-Covid-19 patients with respiratory failure. The investigators also seek to determine the risk factors of these long-term complications in order to guide providers as to which patients should be screened for these deficits. Finally, the investigators will examine the association of various critical care interventions such as invasive versus noninvasive mechanical ventilation or use of sedatives and their effects on disability and cognitive dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* adult patients admitted to the ICU

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients admitted to the intensive care unit
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-04-08 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Life score | up to 12 months after discharge
  SF-36 score

SECONDARY OUTCOMES:
cognitive dysfunction | up to 12 months after discharge
  Montreal Cognitive Assessment (MoCA) score
Functional Status Score | up to 12 months after discharge
  (FSS-ICU)
Physical Disability | up to 12 months after discharge
  MRC neuromuscular Assessment
Psychological Sequelae | up to 12 months after discharge
  Impact Event Score

OTHER OUTCOMES:
hospital anxiety and depression | up to 12 months after discharge
  hospital anxiety and depression scale
ICU related complications | hospitalization up to 6 weeks
  including ventilator associated pneumonia, GI hemorrhage, Deep Vein Thrombosis (DVT) /Pulmonary Embolus (PE), sacral decubitus ulcer, delirium, ICU acquired weakness
hospital discharge location | hospital discharge up to 6 weeks
  measure the location (home, rehabilitation center, nursing home
lCU length of stay | hospitalization up to 6 weeks
  number of days admitted to the ICU
hospital length of stay | hospitalization up to 6 weeks
  number of days admitted to the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No